CLINICAL TRIAL: NCT06109844
Title: FORCEREPAIR - A Wound Exudate Investigation
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Akribes Biomedical GmbH (Unknown); Vascular Research Unit and Department of Vascular Surgery (Unknown)
Responsible Party: Principal Investigator, Frederik Plum, MD, Ph.D Fellow at University of Copenhagen, Bispebjerg Hospital
Other Study IDs: FORCEREPAIR-01; 104834 (Registry Identifier: Research Ethics Comittee)
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Venous Leg Ulcer; Wound Healing; Non-healing Wound; Cytokines
Keywords: Venous Leg Ulcer; Varicose Ulcer; Cytokines; Wound Exudate; Wound Healing; Wound Inflammation; Wound Microbiome
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Wound exudate (twenty-four-hour-collection with Polyurethane foam discs, Bandages, NovaSwab) Tape strips Wound microbiome swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard of Care — Patients enrolled in this observational study receive standard of care. Treatment, ointments, compression and bandages will be registered at every visit.

SUMMARY:
The observational longitudinal study will collect wound exudate from twenty patients with venous leg ulcers. Wound exudate samples are collected using twenty-four-hour collection with polyurethane foam, bandages and the NovaSwab method. Each patient is seen four times where wound exudate and the bacteria microbiome are sampled and wound size is monitored with advanced planimetric tools.

DETAILED DESCRIPTION:
This dual centre longitudinal observational study will run from January 2024 to January 2025. The investigation will include twenty patients over four weeks including four study visits. Sampling of wound exudate can take place on every visit and will be made with the polyurethane discs, the NovaSwab technique and waste bandages. The wound bacteria microbiome is sampled with routine bacterial swabs. Tape strips will be used to assess perilesional skin and control sites of normal skin and will primarily measure skin inflammation parameters. Clinical pictures are taken and analysed using advanced planimetric tools. Patients enrolled receive standard wound care; allowing all kinds of dressing. However when consenting to twenty-four-hour-collection patients will not be allowed to wear active bandages or receive antibiotic treatment for that period. Compression, wound dressings, and use of topical and oral antibiotics will be registered. For the storage of samples, a research biobank is used, and leftover material will be stored in a biobank for future research.

ELIGIBILITY:
Inclusion Criteria:

* Adults fulfilling all inclusion criteria
* Age >18 years
* Venous leg ulcer diagnosis and classic characteristics (localisation, varicose veins, brown-orange hyperpigmentation, leg oedema, stasis dermatitis, atrophie blanche or lipodermatosclerosis) verified by a wound expert (if in doubt venous doppler will be used for verification)
* Wound Area equal to or above 1 cm2 (measured with a ruler length x width)
* Patient can understand Danish
* Patient can comply with protocol
* Patient is fully informed about the study and has given informed consent

Exclusion Criteria:

* Venous leg ulcer with communication to bone
* Known or suspected cancer in the wound
* Allergies towards products used in the study, e.g. polyurethane foam and tegaderm
* Dementia
* Judgement by the investigator that the patient is not suited for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients with venous leg ulcers, verified by a wound expert, will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Wound Exudate Effects on Proliferation of Healthy Primary Human Fibroblasts | Four weeks
  Proliferation
Wound Exudate Effects on Matrix Formation by Healthy Primary Human Fibroblasts | Four weeks
  Matrix Formation
Wound Exudate Effects on Release of Pro-inflammatory Mediators | Four weeks
  Release of pro-inflammatory Mediators
Wound Exudate Effects on Cellular Gene Expression Profiles In Healthy Primary Human Fibroblasts | Four weeks
  Gene Expression Profiles
Exploratory Wound Exudate Compound and Device Testing | Four weeks
  Wound Exudate Compounds

SECONDARY OUTCOMES:
Wound Exudate Profile Relation to Percentage Area Reduction | Four Weeks
Wound Exudate Profile Relation to Wound Microbiome Profile | Four Weeks
Percentage Area Reduction Relation to Wound Microbiome Profile | Four Weeks
Comparisson of Wound Exudate Sampling Techniques | Four Weeks
  Polyurethane disc twenty-four-hour sampling, Bandages and NovaSwabs
Wound Microbiome 16 rRNA/18sRNA | Four Weeks
  Bioburden, Diversity and Pathogens
Wound Perilesional Skin Inflammation | Four Weeks
  Tape Strips from perilesional skin and control site.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Plum, MD, Principal Investigator — Bispebjerg Hospital
Locations (2):
- Denmark (2):
  - Danish Wound Healing Center, Bispebjerg Hospital, Copenhagen, Northwest
  - Vascular Research Unit and Department of Vascular Surgery, Viborg Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data can be shared anonymized upon contact with PI, after publication of primary results.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be avaible after publication of primary results.
Access Criteria: Access upon request via email to Principal Investigator.

REFERENCES:
- [Background] Wolff-Winiski, Barbara, Anton Stütz, and Petra Dörfler. "Methods for identifying a non-healing skin wound and for monitoring the healing of a skin wound." U.S. Patent 11,579,141, issued February 14, 2023
- [Background] Burian EA, Sabah L, Karlsmark T, Kirketerp-Moller K, Moffatt CJ, Thyssen JP, Agren MS. Cytokines and Venous Leg Ulcer Healing-A Systematic Review. Int J Mol Sci. 2022 Jun 10;23(12):6526. doi: 10.3390/ijms23126526. PMID 35742965
- [Background] Serra R, Grande R, Buffone G, Molinari V, Perri P, Perri A, Amato B, Colosimo M, de Franciscis S. Extracellular matrix assessment of infected chronic venous leg ulcers: role of metalloproteinases and inflammatory cytokines. Int Wound J. 2016 Feb;13(1):53-8. doi: 10.1111/iwj.12225. Epub 2014 Feb 19. PMID 24618232
- [Background] Tomic-Canic M, Burgess JL, O'Neill KE, Strbo N, Pastar I. Skin Microbiota and its Interplay with Wound Healing. Am J Clin Dermatol. 2020 Sep;21(Suppl 1):36-43. doi: 10.1007/s40257-020-00536-w. PMID 32914215
- [Background] Versey Z, da Cruz Nizer WS, Russell E, Zigic S, DeZeeuw KG, Marek JE, Overhage J, Cassol E. Biofilm-Innate Immune Interface: Contribution to Chronic Wound Formation. Front Immunol. 2021 Apr 9;12:648554. doi: 10.3389/fimmu.2021.648554. eCollection 2021. PMID 33897696
- [Background] Misic AM, Gardner SE, Grice EA. The Wound Microbiome: Modern Approaches to Examining the Role of Microorganisms in Impaired Chronic Wound Healing. Adv Wound Care (New Rochelle). 2014 Jul 1;3(7):502-510. doi: 10.1089/wound.2012.0397. PMID 25032070
- [Background] Wolcott RD, Hanson JD, Rees EJ, Koenig LD, Phillips CD, Wolcott RA, Cox SB, White JS. Analysis of the chronic wound microbiota of 2,963 patients by 16S rDNA pyrosequencing. Wound Repair Regen. 2016 Jan-Feb;24(1):163-74. doi: 10.1111/wrr.12370. Epub 2015 Dec 10. PMID 26463872
- [Background] Loesche M, Gardner SE, Kalan L, Horwinski J, Zheng Q, Hodkinson BP, Tyldsley AS, Franciscus CL, Hillis SL, Mehta S, Margolis DJ, Grice EA. Temporal Stability in Chronic Wound Microbiota Is Associated With Poor Healing. J Invest Dermatol. 2017 Jan;137(1):237-244. doi: 10.1016/j.jid.2016.08.009. Epub 2016 Aug 24. PMID 27566400
- [Background] Trengove NJ, Bielefeldt-Ohmann H, Stacey MC. Mitogenic activity and cytokine levels in non-healing and healing chronic leg ulcers. Wound Repair Regen. 2000 Jan-Feb;8(1):13-25. doi: 10.1046/j.1524-475x.2000.00013.x. PMID 10760211
- [Background] Wiegand C, Bittenger K, Galiano RD, Driver VR, Gibbons GW. Does noncontact low-frequency ultrasound therapy contribute to wound healing at the molecular level? Wound Repair Regen. 2017 Sep;25(5):871-882. doi: 10.1111/wrr.12595. Epub 2017 Dec 8. PMID 29098740
- [Background] Ambrosch A, Lobmann R, Pott A, Preissler J. Interleukin-6 concentrations in wound fluids rather than serological markers are useful in assessing bacterial triggers of ulcer inflammation. Int Wound J. 2008 Mar;5(1):99-106. doi: 10.1111/j.1742-481X.2007.00347.x. Epub 2008 Jan 3. PMID 18179556
- [Background] Burian EA, Enevold C, Karlsmark T, Agren MS. A simplified method for monitoring cytokines in wound fluid. Wound Repair Regen. 2023 Jan;31(1):47-55. doi: 10.1111/wrr.13053. Epub 2022 Oct 26. PMID 36168150
- See also: FORCE REPAIR website — https://www.forcerepair-wounds.eu/